CLINICAL TRIAL: NCT03760185
Title: Enhanced Pupil Dilation in Patients Taking Alpha-Blockers for Potential Treatment of Intraoperative Floppy Iris Syndrome
Brief Title: Pupil Dilation for Treatment of IFIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-1713
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Intraoperative Floppy Iris Syndrome
MeSH Terms: interventions — Brimonidine Tartrate; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: This is a single arm study in which all enrolled subjects will receive eye drops to only one eye. The alternative eye will serve as the control for efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Brimonidine Tartrate 0.2% (Experimental): One eye was treated with Brimonidine Tartrate 0.2% after a 20-day washout period. Patients will treat right eye 3 times per day for 7 days of treatment.
  Interventions: Drug: Brimonidine Tartrate
- Control - untreated (No Intervention): The left eye will serve as the control for the study and will not receive the Brimonidine Tartrate 0.2% treatment

INTERVENTIONS:
Drug: Brimonidine Tartrate — All subjects will apply brimonidine tartrate to one eye (right eye) only for the duration of study participation.
  Other Names: "Eye Drops"
  Arms: Brimonidine Tartrate 0.2%

SUMMARY:
A novel intervention for targeting the treatment of Intraoperative Floppy Iris Syndrome.

DETAILED DESCRIPTION:
This study explores the effects that medication can have on increasing pupil dilation. Pupil dilation size is important for operative eye procedures. Decreased pupil size is related to increased complication risks in eye surgery. By exploring novel pupil dilation techniques, there is a potential to counteract the effects of poor pupil dilation that is caused by medications such as alpha-blockers. Intraoperative floppy iris syndrome is a syndrome characterized by a floppy iris (IFIS) and poor pupil dilation during surgery that is caused by BPH medications. This study evaluates treatment methods targeting IFIS.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years old or greater) 3. History of having taken, or currently taking any systemic alpha blocker 2. Ability to consent themselves 3. Ability to apply eye drops themselves TID for 7 days

Exclusion Criteria:

1. Subjects with untreated hypertension or baseline BP >160
2. Subjects with Thyrotoxicosis
3. Pregnant women or women trying to conceive
4. Prisoners
5. Inability consent
6. Subjects with anatomical narrow angles or who have never had a dilated eye exam
7. Subjects currently prescribed brimonidine tartrate for glaucoma
8. Subjects who take topical or systemic alpha agonists
9. Patients who take monoamine oxidase (MAO) inhibitors
10. Patients with known severe cardiovascular disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristos Ifantides, MD, Principal Investigator — Denver Health
Locations (1):
- Denver Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be screened at their annual eye examination at the hospital eye clinic.
Units Other Than Participants: eyes
Groups:
- Brimonidine Tartrate 0.2%: All enrolled subjects will receive the interventional drug, Brimonidine tartrate 0.2%, to be applied to ONE eye only.
- Control- Untreated: All subjects enrolled will have one eye serve as a control and will not receive the Brimonidine Tartrate 0.2% treatment
Period: Overall Study
Arm/Group | Brimonidine Tartrate 0.2% | Control- Untreated
Started | 13; 13 eyes | 13; 13 eyes
Completed | 12; 12 eyes | 12; 12 eyes
Not Completed | 1; 1 eyes | 1; 1 eyes
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients in this arm will receive eye drops to be applied to one eye only. The alternative eye will not receive any eye drops and as such will serve as the control.
  Brimonidine Tartrate: All subjects will apply brimonidine tartrate to one eye only for the duration of study participation.
Arm/Group | All Patients
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pre-Study Treatment Pupil Diameter Dilated [Mean (Standard Deviation); unit: milimeters] | 6.50 (1.28)

OUTCOME MEASURES:

1. Primary Outcome: Pupil Dilation Sized of the Treated Eye Compared to the Non-treated Eye
Description: The primary outcome measure is pupil diameter size post dilation (using standard dilating medications of phenylephrine 10%, tropicamide 1%, and cyclopentolate 1%) of the brimonidine tartrate pre-treated eye compared to the non-treated eye
Time Frame: 45 minutes post dilation after 7 days of treatment
Population: One participant did not show for their follow-up visit after treatment.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: eyes
Groups:
- Brimonidine Tartrate 0.2%: The eye that was treated with Brimonidine Tartrate 0.2%.
- Control - Untreated: Eye of participant that was not treated with Brimonidine Tartrate 0.2%
Arm/Group | Brimonidine Tartrate 0.2% | Control - Untreated
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 12 | 12
millimeters | 6.76 (2.57) | 7.17 (1.20)

2. Secondary Outcome: Change in Pupil Diameter of Each Eye After Dilation at the Start of the Study Compared to Pupil Post Dilating Drops at the End of the Study
Description: Change in pupil diameter of each eye after dilation at the start of the study compared to pupil post dilating drops at the end of the study
Time Frame: 45 minutes post dilation after 7 days of treatment
Population: 1 patient did not return for their post-treatment follow-up visit
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: eyes
Groups:
- Brimonidine Tartrate 0.2%: Eye that was treated with Brimonidine Tartrate 0.2%
- Control - Untreated: Eye that was not treated with Brimonidine Tartrate 0.2%
Arm/Group | Brimonidine Tartrate 0.2% | Control - Untreated
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 12 | 12
millimeters | 0.39 (2.20) | 0.91 (1.53)

ADVERSE EVENTS:
Time Frame: up to 30 days from enrollment.
Groups:
- Control- Untreated: The eye that was not treated with Brimonidine Tartrate 0.2%.
Arm/Group | Brimonidine Tartrate 0.2% | Control- Untreated
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/13
Other Adverse Events (participants affected / at risk) | 2/13 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brimonidine Tartrate 0.2% (N=13) | Control- Untreated (N=13)
Surgery- Cryoablation of prostate (Reproductive system and breast disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brimonidine Tartrate 0.2% (N=13) | Control- Untreated (N=13)
Kidney & Urinary tract (Renal and urinary disorders) | 1 (2) | 1 (2)
Ophthalmology - Cataracts (Eye disorders) | 1 (1) | 1 (1)
Cardio - MI (Cardiac disorders) | 1 (1) | 1 (1) — Patient disclosed to study PI that he had an MI and was treated at an outside hospital with a stent surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT03760185/Prot_SAP_002.pdf
  • Informed Consent Form (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03760185/ICF_003.pdf